CLINICAL TRIAL: NCT04876066
Title: Use of Transmucosal Ketamine in Post Stroke Depression
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Amelia Adcock, Associate Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1903509572
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Post-stroke Depression
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: The study will be an open-label study of eligible male and female patients and minorities diagnosed with post stroke depression (PSD) conducted by West Virginia University faculty and research associates.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketamine dose (Experimental): The recommended ketamine dose of 0.5 mg/kg will be administered using a transmucosal route of administration wherein the subject will be instructed to place the liquid solution beneath their tongue and hold it in their mouth for 5 minutes. The pharmacy will prepare two 0.5 mg/kg solutions of ketamine in two syringes for each subject based on subject weight. For example, a 70 kg adult subject will receive a 0.35 mL solution of ketamine. The patient will receive a dose every 7 days for two weeks, for a total of two doses.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Weight-based ketamine dose will be prepared and delivered personally to study physician or study personnel by pharmacy personnel as is done during standard protocol for use of ketamine not part of a clinical study.

SUMMARY:
Studies have shown that ketamine is very effective and has a quick onset in treatment of depression. Most of these studies used intravenous ketamine in an inpatient setting and there are no large trials examining its use in Post Stroke Depression (PSD). There have been only few studies that have used other routes of administration (i.e., oral, transmucosal, intranasal, intramuscular) of ketamine which provided symptom relief for depression. The purpose of this study is to assess the effectiveness and safety of use of transmucosal ketamine in treatment of PSD. We hypothesize that fast acting antidepressant effects can be achieved with tolerable side effects for translation into the general post-stroke population. To test our hypothesis, the specific aim is to: (1) demonstrate that transmucosal administration of ketamine is feasible within the post-stroke depression population and has tolerable side effects. Exploratory aims will include assessment if ketamine also produces fast acting antidepressant effects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (18 years of age or older) of any ethnicity diagnosed with Major Depressive Disorder (DSM-V criteria), who have had failed to respond to prior therapy (as defined as at least one anti-depressant trial or patient was intolerant or noncompliant with anti-depressive medications).
* Willing to take the study drug ketamine on 2 separate occasions and comply with instructions for testing.
* Understands and willing to undergo risks associated with adverse effects of study medications.
* Willing to comply with restrictions and instructions disclosed in the consent form.

Exclusion Criteria:

* Patients with blood pressure over 150 systolic or heart rate over 110 on day of medication administration
* Patients with a diagnosis of epilepsy
* Patients with a significant history of high intraocular pressure.
* Patients with life threatening medical problems.
* Participant is pregnant or breastfeeding.
* Infants and children
* Patients who lack medical decision-making capacity
* Patients who would require medication adjustment during time in the study.
* Known hypersensitivity to the study drug (ketamine).
* Unwilling to undergo risks associated with adverse effects of study drugs.
* Unwilling to comply with restrictions and instructions disclosed in the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms measured by the MADRS. | 14-day dosing period.
  The Montgomery-Asberg Depression Rating Scale is a ten-item diagnostic questionnaire used by mental health clinicians to measure the severity of depressive episodes in subjects with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. "Reduction of MADRS" = 50% drop in total score as compared to baseline, a score of 0-8 indicating NO depression OR a decrease from a more severe category to a more mild one.
Change in depressive symptoms measured by the MADRS-S. | 14-day dosing period.
  Montgomery Asberg Depression Rating Scale Self-assessment (MADRS-S). The overall score ranges from 0-54 with a higher scores indicating more depression.

SECONDARY OUTCOMES:
Side effects will be evaluated using the PRISE. | 14-day dosing period.
  Patient-Rated Inventory of Side Effects (PRISE), perceived tolerance per patient report

CONTACTS AND LOCATIONS:
Locations (1):
- WVU Medicine, Morgantown, West Virginia, United States